CLINICAL TRIAL: NCT06845332
Title: PROTeCt-NEO: Promoting Optimal Treatment Choices Through Implementation of Antibiotic Stewardship Strategies in Neonates With Suspected Early-Onset Sepsis
Brief Title: Promoting Optimal Treatment Choices in Neonates With Suspected Early-Onset Sepsis
Acronym: PrOTeCt-NEO
Status: Recruiting | Type: Observational
Sponsor: Franciscus Gasthuis (Other)
Responsible Party: Sponsor
Other Study IDs: T 110
Record Dates: First submitted 2025-02-18; First posted 2025-02-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Early-onset Sepsis
Keywords: early-onset sepsis; neonatal sepsis; early-onset sepsis calculator; PCT-guided therapy; iv-to-oral switch therapy; implementation
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-implementation cohort
- Post-implementation cohort

SUMMARY:
In this study, three neonatal evidence-based antibiotic stewardship strategies will be implemented in Dutch hospitals. These include the early-onset sepsis (EOS) calculator, procalcitonin (PCT)-guided therapy, and IV-to-oral switch therapy. These strategies have been proven to be effective and safe and are already applied in several Dutch hospitals. However, this is not the case for all hospitals, leading to significant variations in clinical practice. To facilitate the translation of evidence into practice, active implementation will take place.

The primary research design is a prospective implementation study, using a multicenter, non-randomized pre-post design. The aim is to assess the impact of implementing a bundle of antibiotic stewardship interventions (including the EOS calculator, PCT-guided therapy and iv-to-oral switch therapy) in Dutch hospitals, using a multicomponent implementation strategy, on both clinical and implementation outcomes, with a particular focus on evaluating the employed implementation strategies.

A combination of qualitative and quantitative research methods will be used to assess outcomes. Quantitative clinical data from neonates in the pre- and post-implementation periods will be retrospectively collected by the Business Intelligence units of participating hospitals and anonymized before being provided to the central research team. Qualitative data will be gathered through focus groups, interviews, and surveys.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at 34 weeks of gestation or later
* 0-3 days old

Exclusion Criteria:

* stillborn neonates

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population neonates with a minimum postmenstrual age of 34 weeks, between 0-3 days old
Sampling Method: Non-Probability Sample
Enrollment: 55000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Days on therapy | 12 months pre-implementation and 12 months post-implementation

CONTACTS AND LOCATIONS:
Locations (11):
- Netherlands (11):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Gelre Ziekenhuis, Apeldoorn
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Treant Ziekenhuis, Emmen
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Tjongerschans Ziekenhuis, Heerenveen
  - Zuyderland Medisch, Heerlen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Antonius Ziekenhuis Sneek, Sneek

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Achten NB, Klingenberg C, Benitz WE, Stocker M, Schlapbach LJ, Giannoni E, Bokelaar R, Driessen GJA, Brodin P, Uthaya S, van Rossum AMC, Plotz FB. Association of Use of the Neonatal Early-Onset Sepsis Calculator With Reduction in Antibiotic Therapy and Safety: A Systematic Review and Meta-analysis. JAMA Pediatr. 2019 Nov 1;173(11):1032-1040. doi: 10.1001/jamapediatrics.2019.2825. PMID 31479103
- [Background] Keij FM, Kornelisse RF, Hartwig NG, van der Sluijs-Bens J, van Beek RHT, van Driel A, van Rooij LGM, van Dalen-Vink I, Driessen GJA, Kenter S, von Lindern JS, Eijkemans M, Stam-Stigter GM, Qi H, van den Berg MM, Baartmans MGA, van der Meer-Kappelle LH, Meijssen CB, Norbruis OF, Heidema J, van Rossem MC, den Butter PCP, Allegaert K, Reiss IKM, Tramper-Stranders GA. Efficacy and safety of switching from intravenous to oral antibiotics (amoxicillin-clavulanic acid) versus a full course of intravenous antibiotics in neonates with probable bacterial infection (RAIN): a multicentre, randomised, open-label, non-inferiority trial. Lancet Child Adolesc Health. 2022 Nov;6(11):799-809. doi: 10.1016/S2352-4642(22)00245-0. Epub 2022 Sep 9. PMID 36088952
- [Background] Stocker M, van Herk W, El Helou S, Dutta S, Fontana MS, Schuerman FABA, van den Tooren-de Groot RK, Wieringa JW, Janota J, van der Meer-Kappelle LH, Moonen R, Sie SD, de Vries E, Donker AE, Zimmerman U, Schlapbach LJ, de Mol AC, Hoffman-Haringsma A, Roy M, Tomaske M, Kornelisse RF, van Gijsel J, Visser EG, Willemsen SP, van Rossum AMC; NeoPInS Study Group. Procalcitonin-guided decision making for duration of antibiotic therapy in neonates with suspected early-onset sepsis: a multicentre, randomised controlled trial (NeoPIns). Lancet. 2017 Aug 26;390(10097):871-881. doi: 10.1016/S0140-6736(17)31444-7. Epub 2017 Jul 12. PMID 28711318
- [Derived] van Veen LEJ, Tramper-Stranders GA, Achten NB, Plotz FB, van Rossum AMC, Ista E. Implementation strategy for an antibiotic stewardship bundle to promote optimal treatment choices in neonates with suspected early-onset sepsis (Protect-Neo): a study protocol for a multicentre, prospective interrupted time series and before-after study. BMJ Open. 2025 Nov 4;15(11):e103368. doi: 10.1136/bmjopen-2025-103368. PMID 41193205